CLINICAL TRIAL: NCT06408298
Title: A Randomized, Placebo Controlled Proof of Principle (Window of Opportunity) Study of Hydroxychloroquine (HCQ) in Prostate Cancer Patients Undergoing Radical Prostatectomy
Brief Title: HCQ in Resectable Localized Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lionel.D.Lewis, MD (Other)
Collaborators: Dartmouth Cancer Center (Unknown)
Responsible Party: Sponsor-Investigator, Lionel.D.Lewis, MD, Principal Investigator, Professor of Medicine, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 23LEW054|STUDY02002054
Record Dates: First submitted 2024-02-26; First posted 2024-05-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Resectable Localized Prostate Cancer
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): Loading dose 400mg three times a day then 400mg twice daily for up to 28 days prior to surgical resection, taken orally
  Interventions: Drug: Hydroxychloroquine Sulfate 400Mg Tab
- Placebo (Placebo Comparator): Loading dose three times a day then twice daily for up to 28 days prior to surgical resection, taken orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 400Mg Tab — hydroxychloroquine sulfate tablet
  Arms: Hydroxychloroquine
Drug: Placebo — Inactive tablet
  Arms: Placebo

SUMMARY:
This is randomized, double blind, placebo controlled proof of principle (window of opportunity) study of oral hydroxychloroquine in patients with resectable localized prostate cancer. To determine the effects of hydroxychloroquine (HCQ) on markers of autophagy, such as p62, LC3-II and NBR-1 in prostate cancer tissue of patients with resectable localized prostate cancer who undergo radical prostatectomy. To monitor/observe the safety and tolerability of daily oral hydroxychloroquine in the pre and perioperative period in patients who undergo radical prostatectomy. To evaluate the concentration of hydroxychloroquine in normal and prostate tumor tissue and to correlate prostate tissue concentrations with the plasma concentrations in these patients. To perform tumor genomic analysis (for common somatic mutations) and to correlate the molecular response to HCQ and presence/absence of such mutations.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathological confirmation of adenocarcinoma of the prostate Gleason score 6 (grade Group 1) or greater.
* Patients must have resectable prostate cancer as defined by the AJCC (American Joint Committee on Cancer) TNM system and have planned radical prostatectomy.
* Patients must have sufficient tissue from the initial diagnostic prostate biopsy, as determined by the study pathologist, to perform the required study analyses without exhausting the tissue required for clinical purposes
* Age >18 years
* Adequate hematopoietic, hepatic and renal function documented prior to study entry to include: Hb. > 10g/dL, WBC > 3500/mm3, ANC > 1500/mm3 and platelets > 100,000/mm3; hepatic transaminases (AST or ALT) ≤ 2.0 times the upper limits of normal, total bilirubin ≤ 1.5 times the upper limits of normal, estimated creatinine clearance ≥ 60 mL/min or eGFR > 60 mL/min/1.73 m2 and normal serum cations (K+/Mg2+/Ca2+)
* All patients must be medically fit candidates for radical prostatectomy.
* A patient with any retinopathy will only be enrolled into the study with the approval of a board-certified ophthalmologist
* All patients must give informed consent indicating they are aware of the investigational nature of this study treatment prior to any study procedures being performed.

Exclusion Criteria:

* Patients may not have received radiation therapy for their prostate cancer.
* Patients may not have received chemotherapy for their prostate cancer.
* Patients with gastrointestinal abnormalities including: inability to take oral medication, requirement for intravenous alimentation, or prior major surgery or diseases which may cause malabsorption (e.g. bowel resection, ischemic bowel, Crohns or Ulcerative colitis)
* A serious uncontrolled medical disorder or active infection which would impair their ability to receive study treatment will be excluded.
* Patients with significant cardiac disease: including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 3 months, or serious cardiac arrhythmias, including a QT interval corrected for heart rate using the Fridericia formula of ≥ 450 ms, or history of Torsade de pointes will be excluded.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol will be excluded.
* Patients receiving any disease-modifying anti-rheumatic drugs (DMARDs) will be excluded.
* Patients with known or a history of G6PD deficiency will be excluded. Eligible patients will be based on clinician-investigator assessment, that the patient is not at an increased risk for G6PD deficiency (assessment should include information regarding self-reported race/ancestry), OR the patient has a negative screening test for G6PD deficiency.
* Patients taking other commercially available medications which may theoretically either stimulate or inhibit autophagy (calcitriol and chloroquine) will be excluded.
* Patients chronically taking drugs known to cause torsades de pointes will be excluded unless those agents can be discontinued for a period > 6 times their half-life before study enrollment
* Patients with poorly controlled diabetes mellitus will be excluded.
* Patients with a history of epilepsy will be excluded.
* Patients with a history of porphyria will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in expression of markers of autophagy | Day 1, Day 26/27, Day of surgery(approximately day 30)
  To determine the effects of hydroxychloroquine (HCQ) on markers of autophagy, such as p62, LC3-II and NBR-1 in prostate cancer tissue of patients with resectable localized prostate cancer who undergo radical prostatectomy.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 1 through post surgery visit(approximately day 60)
  To monitor/observe the safety and tolerability of daily oral hydroxychloroquine in the pre and perioperative period in patients who undergo radical prostatectomy
Evaluate the concentration of hydroxychloroquine | Day 1, Day 26/27, Day of surgery(approximately day 30)
  To evaluate the concentration of hydroxychloroquine in normal and prostate tumor tissue and to correlate prostate tissue concentrations with the plasma concentrations in these patients.
Measure the tumor mutational burden | Baseline and Day of Surgery(approximately Day 30)
  To perform tumor genomic analysis (for common somatic mutations)
Correlation between tumor mutations and HCQ responses | Baseline and Day of Surgery(approximately Day 30)
  Correlate the molecular response to HCQ and presence/absence of such mutations.

OTHER OUTCOMES:
Exploratory analyses of the effects of hydroxychloroquine on BNIP3 a marker of mitophagy | Baseline and Day of Surgery(approximately Day 30)
  To perform exploratory analyses of the effects of HCQ on the induction of inflammation or necrosis(as measured by BNIP3 expression) in treated as compared to untreated tumors
Explore the effects of hydroxychloroquine on BNIP3 | Baseline and Day of Surgery(approximately Day 30)
  To explore the effects of hydroxychloroquine on BNIP3 expression in prostate cancer tissue

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Lewis, MB BCh., MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans at this time to share IPD